CLINICAL TRIAL: NCT04923113
Title: Comparison of Different Helicobacter Pylori Detection Methods in Patients With Chronic Atrophic Gastritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-0290
Record Dates: First submitted 2021-05-30; First posted 2021-06-11 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2021-05

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — Serologic Tests

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients who meet the inclusion criteria (Experimental): 5 different methods will be performed to detect H. pylori infection in patients who meet the inclusion criteria，and patients with Hp positive will be further treated with 10-day minocycline-based quadruple therapy,to observe the efficacy and safety of minocycline-based regimen for H.pylori eradication as a first-line therapy.
  Interventions: Diagnostic Test: Histology，13C urea breath test，Stool antigen test，Serological antibody test for H.pylori and Serologic test with a current infection marker of H.pylori; Drug: Rabeprazole，Minocycline，Amoxicillin and Colloidal bismuth pectin

INTERVENTIONS:
Diagnostic Test: Histology，13C urea breath test，Stool antigen test，Serological antibody test for H.pylori and Serologic test with a current infection marker of H.pylori — The above 5 detection methods will be performed in patients who meet the inclusion criteria to detect H. pylori infection
Drug: Rabeprazole，Minocycline，Amoxicillin and Colloidal bismuth pectin — Helicobacter pylori positive patients will be treated with rabeprazole10mg,minocycline 100mg,amoxicillin1000mg,and colloidal bismuth pectin 200mg,all twice daily for 10 days

SUMMARY:
As we know，Helicobacter pylori is closely related to many gastrointestinal diseases such as chronic gastritis, peptic ulcer disease,gastric carcinoma and gastric mucosa-associated lymphoid tissue lymphoma，as well as extra-digestive diseases such as urticaria and chronic obstructive pulmonary diseases and so on.The diagnosis of H. pylori infection is based on invasive methods requiring endoscopy and biopsy(e.g. histology, culture, rapid urease test, PCR) or on non-invasive methods (e.g. serology, 13C urea breath test, stool antigen test).Histology has the highest specificity among the others,and also allows us to determine the underlying disease and perform antibiotic sensitivity testing.Serological tests are widely available and more appropriate for epidemiological studies, their main weakness for clinical use is low specificity.The 13C urea breath test is the most accurate method in patients irrespective of age.Stool antigen testing,as a promising method, is easy to perform, and its accuracy may be improved by the use of monoclonal antibodies recently proposed for capturing H. pylori antigen in stool specimen.Sensitivity and specificity, usefulness,and limitation of tests should be considered for selection of detection methods of H. pylori. Our objective is to review the current methods that are used for the detection of H. pylori infection among patients with chronic atrophic gastritis.Except that,patients with Hp positive will be further treated with 10-day minocycline-based quadruple therapy,to observe the efficacy and safety of minocycline-based regimen for H.pylori eradication as a first-line therapy.

DETAILED DESCRIPTION:
Consecutive outpatients (18 to 70 years), with endoscopically proven chronic atrophic gastritis will be enrolled in our study.5 different methods，including histology,13C urea breath test,stool antigen test,serological antibody test for H.pylori and serologic test with a current infection marker of H.pylori，will be performed to detect H. pylori infection.And patients with Hp positive will be further treated with 10-day minocycline-based quadruple therapy.Our objective is to compare specificity and sensitivity of the current methods among patients with chronic atrophic gastritis,meanwhile,to observe the efficacy and safety of minocycline-based regimen for H.pylori eradication as a first-line therapy.

ELIGIBILITY:
Inclusion Criteria:

* participants was confirmed chronic atrophic gastritis by endoscopy
* participants has not been previously received treatment for H.pylori infection.

Exclusion Criteria:

* patients who were allergic to any study medications
* patients who had taken antibiotics,bismuth agent,PPI or H2 receptor antagonist (H2RA) 4 weeks before the study
* patients with previous gastrectomy
* patients with malignancy or severe comorbidity
* pregnant or lactating women
* Patients with poor treatment compliance or could not express themselves correctly
* patients who participated in other drug trial recently (within 3 months of enrollment).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2023-01-18 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of different Helicobacter pylori detection methods | 5 days
  H.pylori infection status will be confirmed by 5 different methods,including histology,13C-UBT,stool antigen test,serological antibody test for H.pylori and serologic test with a current infection marker of H.pylori therapy.

SECONDARY OUTCOMES:
the efficacy of minocycline-based bismuth quadruple therapy for H.pylori eradication as a first-line therapy | 5.5~13.5 weeks
  patients with Hp positive（confirmed by either histology or13C-UBT） will be further treated with 10-day minocycline-based quadruple therapy.The eradication of H.pylori will be confirmed by negative 13C-or 14C-UBT 4~12 weeks after therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Yue-Hua Han, PhD, Study Chair — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- Department of Gastroenterology, The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No